CLINICAL TRIAL: NCT02054455
Title: Protective Effects of Probiotic Administration on SIBO Development and Bowel Symptom Onset in GERD Patients at Long-term PPI Treatment: a Randomized Controlled Cross-sectional Study
Brief Title: Proton Pump Inhibitors and Gastrointestinal Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: University of Catanzaro (Other); Ospedale Nuovo Regina Margherita di Roma Dr. Salvatore Campo (Unknown)
Responsible Party: Principal Investigator, NARDONE GERARDO, ASSOCIATE PROFESSOR OF GASTROENTEROLOGY, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PPI-SIBO-01
Record Dates: First submitted 2012-04-11; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Gastrointestinal Symptoms; Small Intestinal Overgrowth
Keywords: PPI; SIBO; LP-F19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PPI and placebo (Placebo Comparator): Patients will receive PPI and placebo for 3 days/week for 6 months
  Interventions: Dietary Supplement: Placebo
- PPI and Lactobacillus paracasei F19 (Active Comparator): Patients will receive Lactobacillus paracasei F19 in a dose of 25x10E9 live bacterial cells for 3 days/week for 6 months
  Interventions: Dietary Supplement: Lactobacillus paracasei F19
- PPI and Lactobacillus paracasei F19 cross-over 1 (Active Comparator): Patients will receive placebo 3 days/week for the first three months and Lactobacillus paracasei F19 in a dose of 25x10E9 live bacterial cells for 3 days/week for the following three months
  Interventions: Dietary Supplement: Lactobacillus paracasei F19; Dietary Supplement: Placebo
- PPI and Lactobacillus paracasei F19 cross-over 2 (Active Comparator): Patients will receive Lactobacillus paracasei F19 in a dose of 25x10E9 live bacterial cells for 3 days/week for the first three months and placebo 3 days/week for the following three months
  Interventions: Dietary Supplement: Lactobacillus paracasei F19; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei F19 — 25x10E9 live bacterial cells for 3 days/week for 6 months
  Arms: PPI and Lactobacillus paracasei F19; PPI and Lactobacillus paracasei F19 cross-over 1; PPI and Lactobacillus paracasei F19 cross-over 2
Dietary Supplement: Placebo — Placebo will consist of a preparation similar to that of probiotic but with no added microorganisms.
  Arms: PPI and Lactobacillus paracasei F19 cross-over 1; PPI and Lactobacillus paracasei F19 cross-over 2; PPI and placebo

SUMMARY:
The aim of the study is to evaluate the potential protective effect of Lactobacillus paracasei subspecies paracasei F19 administration on bowel symptom onset in patients with gastro-esophageal reflux disease at long-term PPI treatment.

DETAILED DESCRIPTION:
Population and study design

After the approval of the Local Ethical Committee and informed consent of patients, we will consecutively enrol, according to the calculated power of the study, 80 outpatients, among those referred to the Institutional centers on account of recent onset of typical reflux symptoms (heartburn and regurgitation).

Exclusion criteria will be: age <18 or >70 yrs; pregnancy or breast-feeding; evidence of major concomitant diseases (i.e., tumors, cardiovascular disorders and hepatic and/or renal failure); use of PPIs or H2-antagonists, non-steroidal anti-inflammatory drugs (NSAIDs) or antibiotics in the previous 3 months; presence of Helicobacter pylori (H. pylori) infection; erosive esophagitis; presence of bowel symptoms such as bloating, flatulence, abdominal pain, diarrhea and constipation in the last 6 months or irritable bowel syndrome (IBS) according to Rome III criteria.

All patients will undergo upper endoscopy. Patients who will fulfill the entry criteria will be enrolled in the study.

These patients will be treated with pantoprazole 40 mg die for 6 months and they will be randomly assigned to 4 arms:

* the first arm will receive placebo for 3 days/week for 6 months;
* the second arm will receive LP-F19 in a dose of 25x109 live bacterial cells for 3 days/week for 6 months;
* the third arm will receive LP-F19 in a dose of 25x109 live bacterial cells for 3 days/week for the first three months and placebo 3 days/week for the following three months;
* the fourth arm will receive placebo 3 days/week for the first three months and LP-F19 in a dose of 25x109 live bacterial cells for 3 days/week for the following three months.

Placebo will consist of a preparation similar to that of probiotic but with no added microorganisms.

Adherence to treatment Will be evaluated based on self-reporting by the patients and count of returned sackets during monthly control visits. Patients who will take at least 90% of the drugs (pantoprazole, LP-F19 and placebo) for at least 90% of the scheduled time will be considered compliant.

Before starting therapy (i.e. baseline evaluation) and every 4 weeks, each patient will fill up a structured questionnaire for symptom assessment, concerning heartburn and regurgitation, as well as, bowel symptoms, including bloating, abdominal pain, flatulence and bowel habit.

Symptom and bowel habit assessment

Baseline and every 4 weeks after the beginning of the therapy, each patient will fill up a structured questionnaire, focusing on the presence of heartburn, regurgitation, bloating, flatulence, abdominal pain, diarrhea and constipation, with the help of a physician interviewer. The questionnaire, according to a Likert scale, will assess frequency (0 = never, 1 = < 1 episode/week; 2 = < 3 episodes/week; 3 = > 3 episodes/week; 4 = daily episodes) and severity (0 = absent, 1 = mild i.e. not interfering with the daily activities, 2 = moderate i.e. limiting the daily activities, and 3 = severe i.e. hampering the daily activities) of each symptom during the previous 6 months, at baseline and during the last month at every 4-week checkpoints. According to an arbitrary index, symptoms will be considered significant when interfering with daily activities (i.e., mean total score, frequency plus severity, ≥ 4).

Subjects will record their bowel habit on validated diary cards, including every single stool and stool consistency. Stool consistency will be deﬁned according to the Bristol Stool Form Scale (BSFS). Diary cards will be returned every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* recent onset of typical reflux symptoms (heartburn and regurgitation).

Exclusion Criteria:

* age <18 or >70 yrs
* pregnancy or breast-feeding
* evidence of major concomitant diseases (i.e., tumors, cardiovascular disorders and hepatic and/or renal failure)
* use of PPIs or H2-antagonists, non-steroidal anti-inflammatory drugs (NSAIDs) or antibiotics in the previous 3 months
* presence of Helicobacter pylori (H. pylori) infection
* erosive esophagitis
* presence of bowel symptoms such as bloating, flatulence, abdominal pain, diarrhea and constipation in the last 6 months or irritable bowel syndrome (IBS) according to Rome III criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptom's assessment | up to 6 months
  The questionnaire used to assess symptoms was built-up according to a four-point Likert scale evaluating both frequency (0 = never, 1 = < 1 episode/week; 2 = < 3 episodes/week; 3 = > 3 episodes/week; 4 = daily episodes) and severity (0 = absent, 1 = mild i.e. not interfering with the daily activities, 2 = moderate i.e. limiting the daily activities, and 3 = severe i.e. hampering the daily activities) of each symptom during the previous 6 months, at baseline and during the last month at every 4-week checkpoints. According to an arbitrary index, symptoms were considered significant when interfering with daily activities (i.e., mean total score, frequency plus severity, >4).

SECONDARY OUTCOMES:
Bowel habit assessment | up to 6 months
  Subjects will record their bowel habits on validated diary cards, including every single stool and stool consistency. Stool consistency will be deﬁned according to the Bristol Stool Form Scale (BSFS). Diary cards will be returned every four weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University Federico Ii, Naples, Italy